CLINICAL TRIAL: NCT03083054
Title: Cellular Immunotherapy as a Treatment Option for Patients With High Risk Myelodysplastic Syndromes and Acute Myeloid Leukemia
Brief Title: Cellular Immunotherapy for Patients With High Risk Myelodysplastic Syndromes and Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Bruno Deltreggia Benites, Principal Investigator, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1.140.423
Record Dates: First submitted 2017-03-12; First posted 2017-03-17 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): High Risk Myelodysplastic Syndromes or Acute Myeloid Leukemia
  Interventions: Biological: Autologous dendritic cells electroporated with WT1 mRNA

INTERVENTIONS:
Biological: Autologous dendritic cells electroporated with WT1 mRNA — Production and application of autologous dendritic cells vaccines, 4 doses, biweekly

SUMMARY:
The main objective of this work is to conduct a clinical study for the development and application of a vaccine with autologous dendritic cells submitted to electroporation with Wilm's tumor 1 (WT1) messenger ribonucleic acid (mRNA), as an adjuvant treatment of high-risk Myelodysplastic Syndromes and Acute Myeloid Leukemia, aiming to delay the progression of the disease or its relapse and increase overall and event-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18 and 70
* High-risk myelodysplasia (AREB 1 or AREB 2 subtypes) and Acute Myeloid Leukemia
* Minimum interval of 30 days between the last cycle of chemotherapy (when it occurs) and start of immunotherapy
* Performance status between 0 and 3 on the WHO (World Health Organization)-ECOG (Eastern Cooperative Oncology Group) scale
* Calculated creatinine clearance> 30 ml / min using the Cockcroft-Gault formula
* Total bilirubin less than or equal to twice the lower limit of the normal range in the institution and aspartate aminotransferase (AST) less than or equal to twice the upper limit of normal
* Absence of blasts in peripheral blood
* Leukocyte count greater than 3000 cells / mm3, hemoglobin greater than 9.0 g / dl and platelets greater than 70,000 platelets / mm3, if possible. (If the patient does not meet these criteria for apheresis, the possibility of transfusion of blood components after leukapheresis will be proposed and the patient should sign a specific term of science on the possibility of transfusion)
* Normal cardiac evaluation
* Negative serologies for hepatitis B and C viruses and HIV
* Written informed consent form signed before entering the study

Exclusion Criteria:

* Does not meet any of the requirements of the inclusion criteria
* Low risk myelodysplasia by IPSS (International Prognostic Scoring System) or WPSS (WHO adapted Prognostic Scoring System) scores
* Individuals with a history of any previous neoplasia, except those with prolonged clinical remission (more than 5 years) of non-melanoma skin cancers and cervical cancer in situ
* Pregnant or lactating women
* Previous immunotherapy or biological therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology and Transfusion Medicine Center, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No